CLINICAL TRIAL: NCT01344291
Title: Turmeric Effect on Reduction of Serum Prolactin and Related Hormonal Change and Adenoma Size in Prolactinoma Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Haleh Rokni Yazdi, assisstant professor, Mashhad University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Turmeric-01
Record Dates: First submitted 2011-04-18; First posted 2011-04-29 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Hyperprolactinoma
Keywords: hyperprolactinoma; turmeric; amenorrhea
MeSH Terms: conditions — Amenorrhea | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Curcumin — Curcumin is prescribed to new cases of hyperprolactinoma

SUMMARY:
Prolactinoma is the most prevalent anterior hypophysis tumor. The principal treatment for this disorder is Dopamine agonist drugs including bromocriptin and Cabergoline. However, 50% of Bromocriptin treated and 17% of Cabergoline treated patients are resistant to these drugs. Curcumin is the main derivative of turmeric ,an old spice which is used frequently in Indian and Iranian cuisine. It has been proved that curcumin can reduce mammotrope cells proliferation and also intracellular hormone production. The purpose of this study is to evaluate the effect of turmeric on prolactinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* hyperprolactinemia
* microprolactinoma

Exclusion Criteria:

* pregnancy
* macroadenoma
* neurologic signs due to tumor

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
serum prolactin level | 2weeks and one month after treatment

SECONDARY OUTCOMES:
change in LH,FSH and estradiol from baseline | one month ofter treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Mashad University of Medical Sciences, Mashhad, Khorasan Razavi, Iran